CLINICAL TRIAL: NCT04978779
Title: An Open-label, Multicenter Phase 1/1b Study to Characterize Safety, Tolerability, Preliminary Antitumor Activity, Pharmacokinetics, and Pharmacodynamics of VIP152 Monotherapy or Combination Therapy in Subjects With High-risk Chronic Lymphocytic Leukemia or Richter Syndrome
Brief Title: A Study to Evaluate VIP152 in Subjects With Relapsed/Refractory Chronic Lymphocytic Leukemia or Richter Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Vincerx Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VNC-152-102
Record Dates: First submitted 2021-07-15; First posted 2021-07-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Relapsed Non Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; Richter Syndrome; MYC Amplification; MYC Overexpression; MYC Translocation
Keywords: CLL; Leukemia; CDK-9; VIP152; Richter Syndrome; BTKi
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy of VIP152 (Experimental): Investigating VIP152 in a monotherapy cohort in patients with high-risk CLL and Richter Syndrome
  Interventions: Drug: VIP152
- VIP152 in combination with BTKi (Experimental): Investigating VIP152 in combination with a BTKi in patients with CLL
  Interventions: Drug: VIP152; Drug: BTKi

INTERVENTIONS:
Drug: VIP152 — Weekly IV infusion for 28 day cycles.
Drug: BTKi — Taken per local prescribing information
  Arms: VIP152 in combination with BTKi

SUMMARY:
Determine the safety, tolerability, pharmacokinetics, maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of VIP152 as monotherapy or in combination with a BTKi in patients with Chronic Lymphocytic Leukemia (CLL) or Richter Syndrome

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged >/=18 years
* Adequate bone marrow, liver, and renal functions
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Diseases as defined below:

PART1

* Subjects with CLL with either del(17p) by FISH or TP53 mutation who have received ≥1 prior therap(ies) and the last prior regimen must have included venetoclax plus an anti-CD20 antibody and/or a BTKi and did not produce complete remission. Subjects with CLL with either del(17p) by FISH or TP53 mutation who have received ≥2 prior regimens and are intolerant to BTKi and/or venetoclax are also eligible.

or

* Subjects with CLL transformed to DLBCL who have relapsed after, or been refractory, to at least 1 prior line of therapy for DLBCL

PART2

* Subjects with CLL who are currently on an approved BTKi (monotherapy only) at the dose and schedule per the local label for ≥ 12 months who have only achieved SD, PR or PRL

Exclusion Criteria:

* Active clinically serious infections of Grade > 2; requiring parenteral therapy
* Subjects who have new or progressive brain or meningeal or spinal metastases.
* Anticancer chemotherapy or immunotherapy during the study or within one week prior to the first dose of study drug
* Major surgery or significant trauma within 4 weeks before the first dose of study drug
* Allogeneic bone marrow transplant or stem cell rescue within 4 months before first dose of study drug; patients must have completed immunosuppressive therapy before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Up to 3 years
  Number of participants with adverse events as a measure safety and tolerability of high risk CLL and RS in monotherapy

SECONDARY OUTCOMES:
Overall Response Rate | Up to 3 years
  Tumor response evaluation based on the response criteria as applicable for CLL and Richter Syndrome
Duration of Response | Up to 3 years
  Time at Which Response Criteria are Met for Complete Response or Partial Response (Whichever Occurs First) Until the First Date of Recurrence, Progression or Death per applicable response criteria
Progression Free Survival | Up to 3 years
  Number of Participants Without Disease Progression per iwCLL guidelines for CLL & Lugano Classification for NHL
Assessment of pharmacokinetics (PK) of VIP152 | Cycle 1 Day 1 through Cycle 2 Day 1
  Maximum observed drug concentration in measured administration (Cmax) of VIP152
Time To Next Treatment | Up to 3 years
  time from first dose to the initiation of next dose or death

CONTACTS AND LOCATIONS:
Overall Officials: Vincerx Study Director, Study Director — Vincerx Pharma, Inc.
Locations (5):
- United States (4):
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Pratia MCM Krakow, Krakow, Poland

REFERENCES:
- [Derived] Frigault MM, Mithal A, Wong H, Stelte-Ludwig B, Mandava V, Huang X, Birkett J, Johnson AJ, Izumi R, Hamdy A. Enitociclib, a Selective CDK9 Inhibitor, Induces Complete Regression of MYC+ Lymphoma by Downregulation of RNA Polymerase II Mediated Transcription. Cancer Res Commun. 2023 Nov 9;3(11):2268-2279. doi: 10.1158/2767-9764.CRC-23-0219. PMID 37882668